CLINICAL TRIAL: NCT06515509
Title: Evaluation of the Dimensional Alveolar Bone Changes in Immediate Post Extraction Implant Placement in the Maxillary Premolar Area With or Without Loading: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Dimensional Alveolar Bone Changes in Immediate Post Extraction Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Osama Atef Elshahat Attia, Dr. Osama Atef, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-7-23
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Immediate Implant With Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Implants with loading (Active Comparator)
  Interventions: Procedure: immediate implant placement with or without loading
- Immediate Implants without loading (Active Comparator)
  Interventions: Procedure: immediate implant placement with or without loading

INTERVENTIONS:
Procedure: immediate implant placement with or without loading — immediate implant placement with or without loading

SUMMARY:
The aim of this study was to evaluate the dimensional alveolar bone changes in immediate post extraction implant placement with loading compared to immediate post extraction implant placement without loading in the maxillary premolar area . The main question it aims to answer is : Can immediate post extraction implant placement in the maxillary premolar area with loading achieve better alveolar bone dimensions than without loading?

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who have at least one non restorable tooth in the maxillary premolar area that needs to be extracted.

  2. Patients with healthy systemic condition. 3. Patients aged from 20 to 45 years old. 4. Buccal bone thickness should be at least 1mm. (Morton et al., 2014) 5. Availability of bone apical and palatal to the socket to provide primary stability.(Morton et al., 2014) 6. Good oral hygiene.(Wiesner et al., 2010) 7. Accepts one year follow-up period (cooperative patients) Patient provides an informed consent.

  8. Adequate Inter-arch space for implant placement. 9. Favorable occlusion (no traumatic occlusion)

Exclusion Criteria:

- 1. Patients with signs of acute infection related to the area of interest. 2. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits (Lobbezoo et al., 2006).

3. Current and former smokers (Lambert, Morris and Ochi, 2000) 4. Pregnant females.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Height of alveolar bone crest | 6 months
  After the implants are placed, a series of digital radiographs are obtained at 0 , 3, and 6 months duration to study the changes in the amount of crestal bone level.

SECONDARY OUTCOMES:
Implant stability | 6 months
  Implant stability quotient (ISQ) values were measured with an Osstell® (Integration Diagnostics AB, Gothenburg, Sweden)
Alveolar bone width | 6 months
  (CBCT) images are used for evaluation of alveolar bone width around all implant sides all over. At 0. 3, 6 month postoperative by using superimposition and subtraction method
post-surgical patient satisfaction | 6 months
  Post-Surgical Patient Satisfaction Questionnaire (PSPSQ) composed of 3 questions is filled by the patient and numerical score is obtained

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Ekrish AA, Ekram M. A comparative study of the accuracy and reliability of multidetector computed tomography and cone beam computed tomography in the assessment of dental implant site dimensions. Dentomaxillofac Radiol. 2011 Feb;40(2):67-75. doi: 10.1259/dmfr/27546065. PMID 21239568
- [Background] Albrektsson T, Branemark PI, Hansson HA, Lindstrom J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand. 1981;52(2):155-70. doi: 10.3109/17453678108991776. PMID 7246093
- [Background] AlQahtani SM. A novel method of assessment of BMD using CBCT for implant placement: A retrospective study. Medicine (Baltimore). 2023 Jul 7;102(27):e34203. doi: 10.1097/MD.0000000000034203. PMID 37417616
- [Background] Araujo MG, Lindhe J. Ridge alterations following tooth extraction with and without flap elevation: an experimental study in the dog. Clin Oral Implants Res. 2009 Jun;20(6):545-9. doi: 10.1111/j.1600-0501.2008.01703.x. PMID 19515033
- [Background] Atsumi M, Park SH, Wang HL. Methods used to assess implant stability: current status. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):743-54. PMID 17974108
- [Background] Bhola M, Neely AL, Kolhatkar S. Immediate implant placement: clinical decisions, advantages, and disadvantages. J Prosthodont. 2008 Oct;17(7):576-81. doi: 10.1111/j.1532-849X.2008.00359.x. Epub 2008 Aug 26. PMID 18761580
- [Background] Mantena SR, Sivagami G, Gottumukkala SN. Evaluation of crestal bone loss and stability of immediate functional loading versus immediate non-functional loading of single-mandibular posterior implants: A pilot randomized controlled clinical trial. Dent Res J (Isfahan). 2014 Sep;11(5):585-91. PMID 25426151